CLINICAL TRIAL: NCT00175916
Title: An Open-label, Multicenter, Follow-up Trial to Evaluate Long-term Safety and Efficacy of Brivaracetam Used as Adjunctive Treatment at a Flexible Dose up to a Maximum of 200 mg/Day in Subjects Aged 16 Years or Older Suffering From Epilepsy
Brief Title: Follow-up Trial to Evaluate Long-term Safety and Efficacy of Brivaracetam in Subjects Suffering From Epilepsy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N01125; 2004-002140-10 (EudraCT Number)
Expanded Access: NCT03532516 (Available)
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Results first posted 2020-07-16 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Epilepsy
Keywords: Brivaracetam; Epilepsy; long term
MeSH Terms: conditions — Epilepsy | interventions — brivaracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Brivaracetam (Experimental): Flexible dosing, can up and down titrate as needed.
  Interventions: Drug: Brivaracetam (ucb 34714)

INTERVENTIONS:
Drug: Brivaracetam (ucb 34714) — 10 mg and 25 mg tablets. Flexible dosing up to 200 mg/day, twice daily. For each subject, the study will last from study entry until either regulatory approval of brivaracetam has been granted by any Health Authority in an indication of adjunctive treatment of partial onset seizures; or until the Sponsor decides to close the study; until a managed access program, named patient program, compassionate use program, or similar type of access program is established as allowed per country-specific requirements in addition to legal and regulatory guidelines, or until the investigational product development is stopped by the Sponsor.

SUMMARY:
This trial, evaluating the long-term safety and tolerability of brivaracetam, will give subjects suffering from epilepsy, who may have benefited from brivaracetam, the opportunity to continue the treatment. The study will also evaluate the maintenance of efficacy over time of brivaracetam for subjects with partial onset seizures (POS)/primary generalized seizures (PGS).

ELIGIBILITY:
Inclusion Criteria:

* Male/female subjects from 16 years (where legally permitted and ethically accepted) or 18 years onwards suffering from epilepsy and having completed a previous study with brivaracetam as adjunctive treatment, which allowed access to this study
* Subjects with POS/PGS: inpatients or outpatients with epilepsy who participated in previous brivaracetam studies / programs which allow access to the present study
* Subjects with ULD: inpatients or outpatients with epilepsy who were treated with brivaracetam in previous studies / programs which allow access to the present study
* Subjects for whom the Investigator believes a reasonable benefit from the long-term administration of brivaracetam may be expected

Exclusion Criteria:

* Severe medical, neurological and psychiatric disorders, or laboratory values which may have an impact on the safety of the subject
* Poor compliance with visit schedule or medication intake in previous brivaracetam study
* Participation in any clinical study of another investigational drug or device during the study
* Pregnant or lactating woman

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 853 (Actual)
Dates: Start 2005-09 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — +1 844 599 2273 (UCB)
Locations (153):
- United States (3):
  - 935, San Francisco, California
  - 933, Gainesville, Florida
  - 931, Charlottesville, Virginia
- Austria (4):
  - 509, Graz
  - 507, Innsbruck
  - 510, Linz
  - 508, Vienna
- Belgium (6):
  - 501, Edegem, Antwerpen
  - 515, Montignies-sur-Sambre, Chaleroi
  - 506, Bruges
  - 513, Ghent
  - 974, La Louvière
  - 505, Leuven
- Canada (3):
  - 951, Vancouver, British Columbia
  - 950, Montreal, Quebec
  - 952, Québec, Quebec
- Czechia (9):
  - 545, Beroun
  - 543, Brno
  - 544, Brno
  - 546, České Budějovice
  - 519, Ostrava Trebovice
  - 517, Prague
  - 541, Prague
  - 542, Prague
  - 518, Zlín
- Finland (7):
  - 900, Helsinki
  - 581, Kuopio
  - 526, Oulu
  - 582, Oulu
  - 527, Seinäjoki
  - 583, Tampere
  - 811, Tampere
- France (15):
  - 633, Lyon, Bron
  - 632, Angers
  - 628, Béthune
  - 630, Dijon
  - 624, Lille
  - 625, Marseille
  - 623, Montpellier
  - 635, Nancy
  - 626, Paris
  - 920, Paris
  - 622, Rennes
  - 528, Roanne
  - 823, Saint-Pierre-des-Corps
  - 627, Strasbourg
  - 634, Toulouse
- Germany (17):
  - 532, Bad Berka
  - 705, Berlin
  - 708, Berlin
  - 536, Bernau
  - 707, Bielefeld
  - 701, Bonn
  - 709, Erlangen
  - 703, Frankfurt
  - 711, Freiburg im Breisgau
  - 537, Göttingen
  - 535, Jena
  - 710, Kehl
  - 531, Liegau-Augustusbad
  - 533, Mainz
  - 560, München
  - 706, München
  - 704, Ulm
- Hong Kong (2):
  - 649, Hong Kong
  - 650, Shatin
- Hungary (3):
  - 547, Budapest
  - 538, Debrecen
  - 539, Pécs
- 970, Tel Aviv, Israel
- Italy (12):
  - 830, Bologna
  - 553, Foggia
  - 831, Messina
  - 563, Milan
  - 832, Milan
  - 833, Napoli
  - 554, Pavia
  - 550, Perugia
  - 552, Roma
  - 555, Roma
  - 559, Roma
  - 973, Siena
- Netherlands (4):
  - 566, Breda
  - 821, Heemstede
  - 822, Heeze
  - 567, The Hague
- Norway (4):
  - 571, Fredrikstad
  - 568, Oslo
  - 569, Sandvika
  - 570, Trondheim
- Poland (17):
  - 575, Bialystok
  - 741, Gdansk
  - 978, Grodzisk Mazowiecki
  - 748, Katowice
  - 976, Katowice
  - 574, Kielce
  - 975, Krakow
  - 744, Lodz
  - 747, Lodz
  - 742, Lublin
  - 977, Poznan
  - 746, Szczecin
  - 573, Warsaw
  - 576, Warsaw
  - 577, Warsaw
  - 743, Warsaw
  - 745, Warsaw
- Russia (9):
  - 591, Kazan'
  - 578, Moscow
  - 579, Moscow
  - 584, Moscow
  - 586, Moscow
  - 588, Moscow
  - 589, Saint Petersburg
  - 943, Samara
  - 587, Yaroslavl
- Serbia (2):
  - 961, Belgrade
  - 962, Belgrade
- 657, Singapore, Singapore
- 648, George, South Africa
- South Korea (5):
  - 655, Gwangju
  - 652, Seoul
  - 653, Seoul
  - 654, Seoul
  - 656, Seoul
- Spain (8):
  - 599, Alcorcón, Madrid
  - 593, Barcelona
  - 596, Donostia / San Sebastian
  - 594, Madrid
  - 783, Madrid
  - 786, Madrid
  - 595, Vigo
  - 597, Zaragoza
- Sweden (3):
  - 850, Gothenburg
  - 601, Stockholm
  - 604, Umeå
- Switzerland (4):
  - 605, Biel
  - 607, Sankt Gallen
  - 606, Tschugg
  - 608, Zurich
- Taiwan (4):
  - 671, Taichung
  - 672, Taichung
  - 669, Tainan
  - 660, Taoyuan District
- Tunisia (2):
  - 861, Manouba
  - 860, Tunis
- Ukraine (7):
  - 638, Donetsk
  - 637, Kharkiv
  - 641, Kyiv
  - 642, Kyiv
  - 639, Lviv
  - 643, Odesa
  - 640, Uzhhorod

REFERENCES:
- [Result] Moseley BD, Dimova S, Elmoufti S, Laloyaux C, Asadi-Pooya AA. Long-term efficacy and tolerability of adjunctive brivaracetam in adults with focal to bilateral tonic-clonic (secondary generalized) seizures: Post hoc pooled analysis. Epilepsy Res. 2021 Oct;176:106694. doi: 10.1016/j.eplepsyres.2021.106694. Epub 2021 Jun 24. PMID 34218211
- [Derived] Ben-Menachem E, Baulac M, Hong SB, Cleveland JM, Reichel C, Schulz AL, Wagener G, Brandt C. Safety, tolerability, and efficacy of brivaracetam as adjunctive therapy in patients with focal seizures, generalized onset seizures, or Unverricht-Lundborg disease: An open-label, long-term follow-up trial. Epilepsy Res. 2021 Feb;170:106526. doi: 10.1016/j.eplepsyres.2020.106526. Epub 2020 Dec 4. PMID 33461041
- [Derived] Markham A. Brivaracetam: First Global Approval. Drugs. 2016 Mar;76(4):517-22. doi: 10.1007/s40265-016-0555-6. PMID 26899665
- See also: Product Information — http://www.briviact.com/briviact-PI.pdf?v=1479491757
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll patients in September 2005 and concluded in May 2019.
Pre-assignment Details: Participants Flow refers to the Safety Set (SS).
Groups:
- Brivaracetam: Brivaracetam (BRV) was administered with a maximum of 200 mg/day, twice, daily, incremented by 50 mg/day on a weekly basis, during the Up-Titration. During the Down- Titration Period, the BRV dose was decreased in steps of a maximum of 50 mg/day on a weekly basis. A last down-titration step at 20 mg/day for 1 week was included prior to the Post-Treatment Period.
Period: Overall Study
Arm/Group | Brivaracetam
Started | 853
Completed | 234
Not Completed | 619
Not completed — Death | 19
Not completed — Adverse Event | 81
Not completed — Lack of Efficacy | 354
Not completed — Lost to Follow-up | 17
Not completed — Subject Choice | 98
Not completed — Lack of compliance | 8
Not completed — Patient cannot record seizures | 1
Not completed — Sponsor decision | 17
Not completed — Vigabatrin intake | 1
Not completed — Suicidal behaviour | 1
Not completed — Withdrawal by Subject | 1
Not completed — Seizure - free | 4
Not completed — Administrative reason | 1
Not completed — Pregnancy | 1
Not completed — Patient's request | 2
Not completed — Treating physiciant's choice | 1
Not completed — Moved overseas | 1
Not completed — Loss of job and economic burden | 1
Not completed — Site was closed | 9
Not completed — Patient went to prison | 1

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Safety Set which consisted of all participants who took at least 1 dose of study medication.
Arm/Group | Brivaracetam
Number analyzed (Participants) | 853
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14
  Between 18 and 65 years | 827
  >=65 years | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.5 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 418
  Male | 435
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 721
  Black | 2
  Asian | 123
  Other | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least One Treatment-emergent Adverse Event (TEAE)
Description: Treatment-emergent adverse events (TEAEs) were defined as those events which started on or after the date of first dose of investigational medicinal product (IMP), or events in which severity worsened on or after the date of first dose of study medication. The event does not necessarily have a causal relationship with that treatment or usage.
Time Frame: From Entry Visit until Last Visit (up to 162 months)
Population: The Safety Set (SS) consisted of all participants who took at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Groups:
- Brivaracetam (SS): Brivaracetam (BRV) was administered with a maximum of 200 mg/day, twice, daily, incremented by 50 mg/day on a weekly basis, during the Up-Titration. During the Down- Titration Period, the BRV dose was decreased in steps of a maximum of 50 mg/day on a weekly basis. A last down-titration step at 20 mg/day for 1 week was included prior to the Post-Treatment Period. Participants formed the Safety Set (SS).
Arm/Group | Brivaracetam (SS)
Number analyzed (Participants) | 853
Percentage of participants | 84.4

2. Primary Outcome: Percentage of Participants Who Withdrew Due to an Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a participant or trial participant that is administered a drug or biologic (medicinal product) or that is using a medical device. The event does not necessarily have a causal relationship with that treatment or usage.
Time Frame: From Entry Visit until Last Visit (up to 162 months)
Population: The Safety Set (SS) consisted of all participants who took at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Brivaracetam (SS)
Number analyzed (Participants) | 853
Percentage of participants | 11.6

3. Primary Outcome: Percentage of Participants With at Least One Serious Adverse Event (SAE)
Description: A serious adverse event (SAE) is any untoward medical occurrence that at any dose:
  * Results in death
  * Is life-threatening
  * Requires in patient hospitalization or prolongation of existing hospitalization
  * Is a congenital anomaly or birth defect
  * Is an infection that requires treatment parenteral antibiotics
  * Other important medical events which based on medical or scientific judgement may jeopardize the patients or may require medical or surgical intervention to prevent any of the above.
Time Frame: From Entry Visit until Last Visit (up to 162 months)
Population: The Safety Set (SS) consisted of all participants who took at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Brivaracetam (SS)
Number analyzed (Participants) | 853
Percentage of participants | 29.4

4. Secondary Outcome: Partial Onset Seizure (POS) (Type I) Frequency Per 28 Days During the Evaluation Period
Description: The 28 day adjusted seizure frequency was calculated by dividing the number of partial seizures by the number of days for which the diary was completed, and multiplying the resulting value by 28.
  Baseline values for seizure frequency were calculated based on the seizure diary data collected during the baseline period of the previous double-blind studies: N01114 [NCT00175929], N01252 [NCT00490035] and N01254 [NCT00504881].
Time Frame: From Entry Visit until Last Visit (up to 162 months)
Population: The Partial Onset Seizure (POS) Efficacy Analysis Set consisted of all participants with POS who took at least 1 dose of study drug and had at least 1 seizure diary day during the Evaluation Period.
Measure: Median (Inter-Quartile Range); unit: Seizures per 28 days
Groups:
- Brivaracetam (POS Efficacy): Brivaracetam (BRV) was administered with a maximum of 200 mg/day, twice, daily, incremented by 50 mg/day on a weekly basis, during the Up-Titration. During the Down- Titration Period, the BRV dose was decreased in steps of a maximum of 50 mg/day on a weekly basis. A last down-titration step at 20 mg/day for 1 week was included prior to the Post-Treatment Period. Participants formed the Partial Onset Seizure Efficacy Set (POS Efficacy).
Arm/Group | Brivaracetam (POS Efficacy)
Number analyzed (Participants) | 729
Seizures per 28 days
  Baseline | 8.4 [5.0 to 16.1]
  On Treatment | 4.9 [2.1 to 10.8]

5. Secondary Outcome: Percent Change in Partial Onset Seizure (POS) (Type I) Frequency Per 28 Days From Baseline of the Previous Study to the Evaluation Period
Description: The percent change from the previous study baselines, in Partial Onset Seizure (POS) (Type I) frequency per 28 days is defined as:
  (the value at the previous study baselines) minus (the value at each time-points during the evaluation period) divided by the value at the previous study baselines.
  Baseline values for seizure frequency were calculated based on the seizure diary data collected during the baseline period of the previous double-blind studies: N01114 [NCT00175929], N01252 [NCT00490035] and N01254 [NCT00504881].
Time Frame: From Entry Visit until Last Visit (up to 162 months)
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Brivaracetam (POS Efficacy)
Number analyzed (Participants) | 729
Percent change | 43.1 [9.9 to 71.5]

6. Secondary Outcome: Responder Rate in POS (Type I) Frequency Over the Evaluation Period
Description: A responder is defined as a participant with a ≥ 50% reduction in seizure frequency from the Baseline Period of the previous study.
  Baseline values for seizure frequency were calculated based on the seizure diary data collected during the baseline period of the previous double-blind studies: N01114 [NCT00175929], N01252 [NCT00490035] and N01254 [NCT00504881].
Time Frame: From Entry Visit until Last Visit (up to 162 months)
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Brivaracetam (POS Efficacy)
Number analyzed (Participants) | 729
Percentage of participants | 43.6

ADVERSE EVENTS:
Time Frame: From Entry Visit until Last Visit (up to 162 months)
Arm/Group | Brivaracetam (SS)
All-Cause Mortality (participants affected / at risk) | 19/853
Serious Adverse Events (participants affected / at risk) | 248/853
Other Adverse Events (participants affected / at risk) | 569/853
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brivaracetam (SS) (N=853)
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 2 (2)
Acute coronary syndrome (Cardiac disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1)
Cardiac disorder (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Baltic myoclonic epilepsy (Congenital, familial and genetic disorders) | 2 (5)
Vertigo (Ear and labyrinth disorders) | 4 (6)
Hypoacusis (Ear and labyrinth disorders) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Thyroiditis (Endocrine disorders) | 1 (1)
Cataract (Eye disorders) | 2 (2)
Corneal erosion (Eye disorders) | 1 (1)
Opsoclonus myoclonus (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Visual impairment (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 5 (5)
Vomiting (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (4)
Dysphagia (Gastrointestinal disorders) | 2 (4)
Gastric ulcer (Gastrointestinal disorders) | 2 (2)
Gastritis (Gastrointestinal disorders) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Abdominal hernia (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1)
Duodenitis (Gastrointestinal disorders) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1)
Gastric polyps (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (3)
Intestinal obstruction (Gastrointestinal disorders) | 1 (4)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Proctocolitis (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 5 (5)
Death (General disorders) | 4 (4)
Fatigue (General disorders) | 2 (2)
Unevaluable event (General disorders) | 2 (4)
Chest pain (General disorders) | 1 (1)
Device failure (General disorders) | 1 (1)
Drowning (General disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Haemorrhagic cyst (General disorders) | 1 (1)
Implant site haematoma (General disorders) | 1 (1)
Irritability (General disorders) | 1 (1)
Sudden death (General disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 3 (3)
Biliary colic (Hepatobiliary disorders) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1)
Immunodeficiency (Immune system disorders) | 1 (1)
Pneumonia (Infections and infestations) | 9 (14)
Sepsis (Infections and infestations) | 6 (6)
Upper respiratory tract infection (Infections and infestations) | 4 (4)
Urinary tract infection (Infections and infestations) | 4 (4)
Appendicitis (Infections and infestations) | 2 (2)
Postoperative wound infection (Infections and infestations) | 2 (2)
Pyelonephritis (Infections and infestations) | 2 (2)
Septic shock (Infections and infestations) | 2 (2)
Skin infection (Infections and infestations) | 2 (2)
Bronchitis (Infections and infestations) | 1 (1)
Bronchopneumonia (Infections and infestations) | 1 (2)
Device related infection (Infections and infestations) | 1 (1)
Ear infection (Infections and infestations) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Incision site infection (Infections and infestations) | 1 (1)
Infected bites (Infections and infestations) | 1 (1)
Localised infection (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Pneumonia mycoplasmal (Infections and infestations) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Tuberculosis (Infections and infestations) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1)
Vestibular neuronitis (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 10 (11)
Clavicle fracture (Injury, poisoning and procedural complications) | 5 (5)
Contusion (Injury, poisoning and procedural complications) | 5 (5)
Ankle fracture (Injury, poisoning and procedural complications) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 4 (8)
Femur fracture (Injury, poisoning and procedural complications) | 4 (4)
Laceration (Injury, poisoning and procedural complications) | 4 (4)
Concussion (Injury, poisoning and procedural complications) | 3 (3)
Extradural haematoma (Injury, poisoning and procedural complications) | 3 (3)
Facial bones fracture (Injury, poisoning and procedural complications) | 3 (3)
Hand fracture (Injury, poisoning and procedural complications) | 3 (3)
Spinal fracture (Injury, poisoning and procedural complications) | 3 (3)
Toxicity to various agents (Injury, poisoning and procedural complications) | 3 (3)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2)
Jaw fracture (Injury, poisoning and procedural complications) | 2 (2)
Ligament rupture (Injury, poisoning and procedural complications) | 2 (2)
Lower limb fracture (Injury, poisoning and procedural complications) | 2 (2)
Meniscus lesion (Injury, poisoning and procedural complications) | 2 (2)
Poisoning (Injury, poisoning and procedural complications) | 2 (2)
Skull fracture (Injury, poisoning and procedural complications) | 2 (2)
Skull fractured base (Injury, poisoning and procedural complications) | 2 (2)
Thermal burn (Injury, poisoning and procedural complications) | 2 (2)
Tibia fracture (Injury, poisoning and procedural complications) | 2 (2)
Upper limb fracture (Injury, poisoning and procedural complications) | 2 (2)
Accident (Injury, poisoning and procedural complications) | 1 (1)
Accidental exposure (Injury, poisoning and procedural complications) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1)
Bursa injury (Injury, poisoning and procedural complications) | 1 (1)
Cartilage injury (Injury, poisoning and procedural complications) | 1 (1)
Chest injury (Injury, poisoning and procedural complications) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Incorrect dose administered (Injury, poisoning and procedural complications) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Muscle rupture (Injury, poisoning and procedural complications) | 1 (1)
Near drowning (Injury, poisoning and procedural complications) | 1 (1)
Open wound (Injury, poisoning and procedural complications) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1)
Postoperative hernia (Injury, poisoning and procedural complications) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Spinal column injury (Injury, poisoning and procedural complications) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1)
Investigation (Investigations) | 1 (1)
Thyroid function test abnormal (Investigations) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 6 (6)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Histamine intolerance (Metabolism and nutrition disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 7 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 2 (2)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Femoroacetabular impingement (Musculoskeletal and connective tissue disorders) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4)
Astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ependymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Mixed oligo-astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Testicular neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Convulsion (Nervous system disorders) | 36 (54)
Epilepsy (Nervous system disorders) | 11 (13)
Status epilepticus (Nervous system disorders) | 10 (12)
Grand mal convulsion (Nervous system disorders) | 8 (12)
Myoclonus (Nervous system disorders) | 9 (20)
Myoclonic epilepsy (Nervous system disorders) | 4 (11)
Seizure cluster (Nervous system disorders) | 4 (4)
Somnolence (Nervous system disorders) | 3 (3)
Cerebrovascular accident (Nervous system disorders) | 2 (2)
Complex partial seizures (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 2 (2)
Partial seizures with secondary generalisation (Nervous system disorders) | 2 (2)
Altered state of consciousness (Nervous system disorders) | 1 (1)
Ataxia (Nervous system disorders) | 1 (2)
Aura (Nervous system disorders) | 1 (1)
Balance disorder (Nervous system disorders) | 1 (1)
Brachial plexopathy (Nervous system disorders) | 1 (1)
Cerebral haematoma (Nervous system disorders) | 1 (2)
Cerebral infarction (Nervous system disorders) | 1 (1)
Coordination abnormal (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1)
Encephalitis (Nervous system disorders) | 1 (1)
Hemiplegia (Nervous system disorders) | 1 (1)
Hydrocephalus (Nervous system disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
Partial seizures (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Psychomotor hyperactivity (Nervous system disorders) | 1 (1)
Radiculitis lumbosacral (Nervous system disorders) | 1 (1)
Status migrainosus (Nervous system disorders) | 1 (2)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1)
Toxic encephalopathy (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 4 (4)
Abortion (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Abortion complete (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Foetal growth restriction (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Pregnancy on contraceptive (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Pregnancy on oral contraceptive (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 7 (7)
Depression (Psychiatric disorders) | 6 (7)
Psychotic disorder (Psychiatric disorders) | 3 (4)
Aggression (Psychiatric disorders) | 3 (3)
Suicide attempt (Psychiatric disorders) | 3 (3)
Abnormal behaviour (Psychiatric disorders) | 2 (2)
Acute psychosis (Psychiatric disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 2 (2)
Confusional state (Psychiatric disorders) | 2 (2)
Depressed mood (Psychiatric disorders) | 2 (2)
Dysthymic disorder (Psychiatric disorders) | 2 (2)
Suicidal behaviour (Psychiatric disorders) | 2 (2)
Agitation (Psychiatric disorders) | 1 (1)
Conversion disorder (Psychiatric disorders) | 1 (2)
Decreased interest (Psychiatric disorders) | 1 (1)
Delirium tremens (Psychiatric disorders) | 1 (1)
Dissociative disorder (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Mental disorder (Psychiatric disorders) | 1 (4)
Panic attack (Psychiatric disorders) | 1 (1)
Panic disorder (Psychiatric disorders) | 1 (1)
Polydipsia psychogenic (Psychiatric disorders) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 3 (6)
Bladder pain (Renal and urinary disorders) | 1 (1)
Calculus bladder (Renal and urinary disorders) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 1 (1)
Calculus urinary (Renal and urinary disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1)
Urinary tract disorder (Renal and urinary disorders) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 4 (4)
Epididymitis (Reproductive system and breast disorders) | 1 (1)
Menometrorrhagia (Reproductive system and breast disorders) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1)
Menstrual disorder (Reproductive system and breast disorders) | 1 (1)
Pelvic fluid collection (Reproductive system and breast disorders) | 1 (1)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatomyositis (Skin and subcutaneous tissue disorders) | 1 (1)
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1)
Artificial urinary sphincter implant (Surgical and medical procedures) | 1 (1)
Cataract operation (Surgical and medical procedures) | 1 (1)
Cholecystectomy (Surgical and medical procedures) | 1 (1)
Gallbladder operation (Surgical and medical procedures) | 1 (1)
Hernia repair (Surgical and medical procedures) | 1 (1)
Radiotherapy (Surgical and medical procedures) | 1 (1)
Shoulder operation (Surgical and medical procedures) | 1 (1)
Tonsillectomy (Surgical and medical procedures) | 1 (1)
Tracheostomy (Surgical and medical procedures) | 1 (1)
Urethral repair (Surgical and medical procedures) | 1 (1)
Circulatory collapse (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1)
Venous thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brivaracetam (SS) (N=853)
Vertigo (Ear and labyrinth disorders) | 58 (114)
Diarrhoea (Gastrointestinal disorders) | 78 (112)
Nausea (Gastrointestinal disorders) | 55 (78)
Vomiting (Gastrointestinal disorders) | 53 (89)
Fatigue (General disorders) | 84 (106)
Nasopharyngitis (Infections and infestations) | 157 (332)
Urinary tract infection (Infections and infestations) | 75 (125)
Influenza (Infections and infestations) | 66 (104)
Upper respiratory tract infection (Infections and infestations) | 50 (127)
Bronchitis (Infections and infestations) | 47 (68)
Fall (Injury, poisoning and procedural complications) | 47 (62)
Contusion (Injury, poisoning and procedural complications) | 45 (68)
Back pain (Musculoskeletal and connective tissue disorders) | 77 (99)
Arthralgia (Musculoskeletal and connective tissue disorders) | 52 (73)
Headache (Nervous system disorders) | 186 (419)
Dizziness (Nervous system disorders) | 123 (191)
Convulsion (Nervous system disorders) | 112 (158)
Somnolence (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 73 (104)
Insomnia (Psychiatric disorders) | 71 (95)
Depression (Psychiatric disorders) | 65 (80)
Hypertension (Vascular disorders) | 43 (53)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2015-03-12): https://cdn.clinicaltrials.gov/large-docs/16/NCT00175916/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-11): https://cdn.clinicaltrials.gov/large-docs/16/NCT00175916/SAP_001.pdf